CLINICAL TRIAL: NCT02215850
Title: A Phase I, Multi-center, Open-label, Study to Investigate the Safety, Tolerability and Pharmacokinetic of SLC-0111 in Subjects With Advanced Solid Tumours
Brief Title: Safety Study of SLC-0111 in Subjects With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Welichem Biotech Inc. (Industry)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-055/SLC0111-14-C01
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Solid Tumours
MeSH Terms: interventions — SLC-0111

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SLC-0111 (Experimental)
  Interventions: Drug: SLC-0111

INTERVENTIONS:
Drug: SLC-0111

SUMMARY:
SLC-0111 is a selective, small molecule, inhibitor of carbonic anhydrase (CA) IX and is in development for the treatment of solid tumours over-expressing CA IX. CAIX, a transmembrane metalloenzyme, is overexpressed on extracellular surfaces of hypoxic tumour cells but its expression is highly restricted in normal tissue. CAIX is a functional regulator of processes critical for tumour growth and metastasis, including pH regulation, survival, migration and invasion.

This prospective single arm study will evaluate the safety of SLC-0111 given once daily in 28 day cycles in subjects with advanced solid tumours. The intent of this research study is to find our more information such as: the highest dose of SLC-0111 that can be given safely, the side effect it may cause, to examine how the body affects the study drug concentration in the blood (pharmacokinetics or PK), and to gain some information on its effectiveness in treating cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years old.
2. Able and willing to provide written informed consent and to comply with the study protocol and procedures.
3. Histological or cytological evidence of advanced and/or metastatic or unresectable tumour(s) for which standard curative measures do not exist.
4. Recovery to ≤ Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Life expectancy greater than 3 months in the Investigator's opinion.
7. The following time must have elapsed between previous therapy for cancer and first administration of SLC-0111:

   * At least 4 weeks since previous cancer-directed therapy (cytotoxic agents, targeted therapy including monoclonal antibody therapy, immunotherapy, hormonal therapy, and prior radiotherapy).
   * At least 4 weeks or five times the elimination half-life (whichever is shortest) of any investigational drug/biologic or combination product prior to first dose of study treatment.
   * At least 3 months since prior interferon therapy.
   * At least 4 weeks since any major surgery
   * At least 12 weeks since any incidence of severe gastrointestinal bleeding.
8. Adequate renal function:

   • Creatinine ≤1.5 times upper limit of normal (ULN) or calculated creatinine clearance (CrCl) using the Cockcroft Gault formula ≥60 mL/min, or measured CrCl ≥60 mL/min.
9. Adequate hepatic function:

   * Serum bilirubin ≤1.5 times upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (≤5 x ULN if liver lesions present [i.e. liver metastasis or primary tumour of the liver for hepatocellular carcinoma (HCC]).
10. Adequate bone marrow function:

    * Absolute neutrophil count ≥1.5 x 109/L
    * Platelets ≥100 x 109/L
    * Haemoglobin ≥90 g/L
11. Adequate coagulation tests: international normalised ratio (INR) ≤1.5 x ULN.
12. Corrected QT interval (QTcB) < 470 ms
13. Ability to take oral liquid medication
14. Negative urine pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential, defined as a sexually mature woman who has not undergone a hysterectomy/oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months).
15. Sexually-active women of child-bearing potential and sexually-active male subjects with a female partner of child-bearing potential or pregnant must agree to use acceptable double-barrier methods of contraception to avoid pregnancy from screening, for the duration of the study, and for 4 months after the last dose of study drug (Rhythm methods and/or abstinence will not be considered as highly effective methods of birth control).
16. Subjects must agree not to donate gametes (i.e. sperms and eggs) during the study and for 4 months following their last dose of SLC-0111.

Exclusion Criteria:

1. Prior treatment with any drugs known to inhibit hypoxia (drugs that function under hypoxia and drugs that target cells in hypoxic regions are allowed).
2. Females who are pregnant, planning to become pregnant or breastfeeding.
3. Known central nervous system metastasis that is symptomatic and/or requires treatment. Radiographically stable lesions for 3 months prior to enrollment that were previously treated with steroids are permitted as long as they are not currently being treated with steroids.
4. History of myocardial infarction, unstable angina, congestive heart failure (New York Heart Association class III/IV), cerebrovascular accident, transient ischaemic attack, limb claudication at rest in the 6 months prior to the first administration of SLC-0111, or ongoing symptomatic dysrhythmias, or uncontrolled atrial or ventricular arrhythmias, or uncontrolled hypertension defined as systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg, or left ventricular ejection fraction (LVEF) <50%.
5. Any condition or illness that, in the opinion of the Investigator would compromise subject safety or interfere with the evaluation of the safety of the study drug.
6. Subjects with documented cases of human immunodeficiency virus (HIV), or hepatitis B or C.
7. Concurrent treatment with warfarin (Coumadin).
8. Known allergy to study drug or its excipients (PEG 200, PEG 400, Soy lecithin, Vitamin E TPGS, and Propylene glycol) or severe allergy to other sulfonamides.
9. Gastrointestinal condition which could interfere with the swallowing or absorption of study medication.
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, gastrointestinal bleeding, ulceration, or perforation within 12 weeks prior to the first administration of SLC-0111 or significant bowel resection that would preclude adequate absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 year. Subjects will continue to receive SLC-0111 for multiple cycles of 28 days if they are receiving benefit from therapy.
  To evaluate the safety and tolerability of SLC-0111, administered once daily, in subjects with advanced solid tumours.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SLC-0111 | 1 year.
  Changes in AUC over time in subjects taking SLC-0111 once daily.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Alberta Health Services - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario